CLINICAL TRIAL: NCT05184790
Title: LEARN: Learning Environment for Artificial Intelligence in Radiotherapy New Technology
Acronym: LEARN
Status: Recruiting | Type: Observational
Sponsor: University of Sydney (Other)
Collaborators: Princess Alexandra Hospital, Brisbane, Australia (Other); Calvary Mater Newcastle, Australia (Other); Western Sydney Local Health District (Other); Austin Health (Other Government); Peter MacCallum Cancer Centre, Australia (Other)
Responsible Party: Sponsor
Other Study IDs: IX-2021-DS-LEARN
Record Dates: First submitted 2021-12-22; First posted 2022-01-11 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Arrhythmias, Cardiac; Breast Cancer; Prostatic Cancer; Brain Cancer; Kidney Cancer; Head and Neck Cancer; Liver Cancer; Pancreatic Cancer; Spinal Neoplasm
Keywords: Radiation Therapy; markerless tracking
MeSH Terms: conditions — Arrhythmias, Cardiac; Breast Neoplasms; Prostatic Neoplasms; Brain Neoplasms; Kidney Neoplasms; Head and Neck Neoplasms; Liver Neoplasms; Pancreatic Neoplasms; Spinal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (9):
- Brain cancer: Patients having radiation therapy for treatment of brain cancer.
- Breast cancer: Patients having radiation therapy for treatment of breast cancer.
- Head and neck cancer: Patients having radiation therapy for treatment of head and neck cancer.
- Kidney cancer: Patients having radiation therapy for treatment of kidney cancer.
- Liver cancer: Patients having radiation therapy for treatment of liver cancer.
- Pancreatic cancer: Patients having radiation therapy for treatment of pancreatic cancer.
- Prostatic cancer: Patients having radiation therapy for treatment of prostate cancer.
- Spinal neoplasm: Patients having radiation therapy for treatment of spinal cancer.
- Cardiac arrhythmia: Patients having radiation therapy for treatment of cardiac arrhythmia

SUMMARY:
This study will develop a whole-of-body markerless tracking method for measuring the motion of the tumour and surrounding organs during radiation therapy to enable real-time image guidance.

Routinely acquired patient data will be used to improve the training, testing and accuracy of a whole-of-body markerless tracking method. When the markerless tracking method is sufficiently advanced, according to the PI of each of the data collection sites, the markerless tracking method will be run in parallel to, but not intervening with, patient treatments during data acquisition.

DETAILED DESCRIPTION:
This observational study will access routinely acquired radiation therapy treatment data from 300 patients including brain, breast, head and neck, kidney, liver, pancreas, prostate, spine and cardiac anatomic sites. At least 30 patients will be recruited from each anatomic site to enable sufficient data for the markerless tracking method training, testing and validation. The clinical data will be used to develop, train, test and validate a markerless target tracking method.

After the treatment, the ground truth and the variability in the ground truth will be computed. The patient images, the markerless tracking results, the ground truth and the variability will be uploaded to an in-house developed clinical trial learning system. Uploading additional data to the learning system automatically triggers the model building of the deep learning system. In this manner, the learning system gets both more accurate and more robust with each patient accrued. As the patient data accrues, the primary hypothesis of targeting accuracy can be tested.

The developed markerless tracking software will be applied by study personnel to the treatment imaging data for each anatomic site using five-fold cross-validation where 80% of the data is used for training and the remaining unseen 20% of the data is used for testing. Target positions produced by the markerless tracking will be compared with a 'ground truth'.

ELIGIBILITY:
Inclusion Criteria:

* Will receive radiation therapy for brain, breast, head and neck, kidney, liver, pancreas, prostate, spine cancer treatment or cardiac arrhythmia treatment at a participating centre.
* Will receive CT planning, and a cone beam CT scan for at least one fraction of radiation therapy.
* Will receive intrafraction x-ray imaging for the liver, pancreas, prostate, spine cancer treatment or cardiac arrhythmia treatment. As intrafraction imaging is not common standard of care for brain, breast, head and neck and kidney cancer treatments there is no requirement to have intrafraction x-ray imaging data for these anatomical sites.
* Provides written informed consent.

Exclusion Criteria:

* Less than 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 300 participants, at least 30 from each of nine cohorts of anatomical sites receiving radiation therapy treatment.
  Eight cohorts include: those being treated for cancer at anatomical sites of brain, head and neck, breast, liver, pancreas, kidney, prostate, spine; those being treated for cardiac arrhythmia.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-02-28 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Accuracy of markerless tracking | 3 years
  Proportion of markerless tracking within 5 mm of the ground truth for each of nine anatomical sites (cohorts)

SECONDARY OUTCOMES:
Clinical acceptability of markerless tracking system | 3 years
  Proportion of radiation therapists considering the markerless tracking system acceptable using a survey

CONTACTS AND LOCATIONS:
Overall Officials: Paul Keall, Study Chair — Professor
Locations (4):
- Australia (4):
  - Royal North Shore Hospital, Saint Leonards, New South Wales
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Alfred Health, Melbourne, Victoria
  - Peter MacCallum Cancer Centre, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: Yes
After study completion, de-identified (non-coded, non-re-identifiable) data will be available to researchers for further scientific research. Information about data sharing will be provided to study participants in the Patient Information Sheet.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After study completion.
Access Criteria: Data stored at the university: In order to download / decompress the stored, de-identified data, participating researchers will agree to the terms of use for the data, including that the data are not to be published or otherwise redistributed without the express consent of the original investigator(s).
  Data stored at an external repository: de-identified study data may be provided to an external research data repository, archive or register so that it may be made publicly available for other scientific research. Study data that are provided to an external research data repository will be stored at and managed by the external repository. Data will only be shared with repositories whose function has been reviewed and approved by an accredited Research Integrity/Ethics Committee/Board, under a Materials Transfer Agreement with the University.